CLINICAL TRIAL: NCT03488134
Title: A Prospective Study of Predicting Prognosis and Recurrence of Thyroid Cancer Via New Biomarkers, Urinary Exosomal Thyroglobulin and Galectin-3
Brief Title: Predicting Prognosis and Recurrence of Thyroid Cancer Via New Biomarkers, Urinary Exosomal Thyroglobulin and Galectin-3
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201711082RINA
Record Dates: First submitted 2018-03-28; First posted 2018-04-04 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Thyroid Cancer
Keywords: Exosome; Anaplastic thyroid cancer; Urine; Biological marker; Thyroglobuin; Galectin-3
MeSH Terms: conditions — Thyroid Neoplasms; Thyroid Carcinoma, Anaplastic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Although thyroid cancers are low-grade endocrine malignancy, most patients usually received thyroidectomy with ablative radioactive iodine therapy. Such patients were followed with thyroid ultrasonography and serial serum thyroglobulin evaluation. Prior researches indicated that one-third well-differentiated thyroid cancers could transform to poorly-differentiated patterns, even to be anaplastic thyroid cancer (ATC), a fatal malignancy, and no effective therapeutic strategies was noted, including surgical intervention, chemotherapy and radiotherapy. The poorly-differentiated or anaplastic change of thyroid cancer cells proliferates rapidly and always invades local tissues with distant metastasis. Cellular de-differentiation is the most pivotal cause for malignant transformation and invasion. De-differentiation usually in papillary thyroid cancer and follicular thyroid cancer, and definitely in ATC. Therefore, the investigators try to find the biological markers and therapeutic targets via the exosomal expression in urine. On the continuing basis of prior ATC cells culture experiments.

Exosomes are nanovesicles secreted into extracellular environments. Cancer cell-derived exosomes could be found in plasma, saliva, urine and other body fluid of patients with cancer. The investigators try to analyze the urinary exosomal proteins, including thyroglobulin and galectin-3, to find the early prognostic biological markers in urine via this prospective study.

The investigators expected to enroll 150 post-operative patients with papillary, follicular or anaplastic thyroid cancer, and collect the urine samples in outpatient clinic per year. The investigators will analyze the urine exosomal proteins and probable biological markers, including thyroglobulin and galectin-3. The investigators hope to find the prognostic biological markers via this prospective study. The investigators further hope to find newly therapeutic and follow-up pathway for such patients with well-differentiated or anaplastic thyroid cancer.

DETAILED DESCRIPTION:
Papillary and follicular thyroid cancers are low-grade endocrine malignancy, and most patients usually received thyroidectomy with ablative radioactive iodine therapy. These patients were followed with thyroid ultrasonography and serial serum thyroglobulin evaluation. Serum thyroglobulin is the pivotal biomarker in survey of possible residual tumor or recurrence of thyroid cancer. Generally, such patients appear to have the higher residual risk of isolated thyroglobulinemia, and postoperative serum thyroglobulin may suggest distant metastases. Low-risk patients with a non-stimulated postoperative serum thyroglobulin was usually defined of less than 0.4 ng/mL or with thyroid hormone withdrawal thyroglobulin of less than 1.0 ng/mL. However, expensive recombinant human TSH (rhTSH) is usually needed to stimulate serum thyroglobulin for detecting local recurrence or distant metastasis. The issue of earlier biological markers for predicting prognosis of thyroid cancer should be raised.

Exosomes are nanovesicles secreted into extracellular environments. Cancer cell-derived exosomes could be found in plasma, saliva, urine and other body fluid of patients with cancer. A growing evidence suggests that exosomes could be used as biomarkers to be the diagnosis and prognosis of malignant tumors. Exosomes are 40-100 nm diameters, and correspond to the intraluminal vesicles of endosomal multivesicular bodies. Exosomes secreted by cells could micro-molecularly transfer messages between cells, and be the biological markers of cancer. In addition, exosomes could be collected in serum, tissue fluid and urine for diseases follow-up, and urine as the biosample is easier to repeatedly obtain and non-invasive. In this study, the investigators enroll patients with papillary, follicular, and collect the urine samples before operation, immediately after operation, post-operatively. The investigators try to analyze the urinary exosomal proteins to find the early prognostic biological markers in urine via this prospective study.

This pilot study report will explore that urinary exosomal thyroglobulin could be a reliable biological marker to substitute for serum thyroglobulin in the future. Such patient do not need to withdraw thyroid hormone or receive rhTSH stimulation. For patients with thyroid cancer, if they received thyroidectomy with ablative radioactive I-131 therapy, serum thyroglobulin is defined to be cancer biomarker in the course of follow-up. If thyroglobulin cannot be detected in serum, then such patients were suggested to be biochemically complete treatment, independent of the interference of anti-thyroglobulin antibody. Usually, serum thyroglobulin cannot be detected even under expensive rhTSH stimulation in patients of biochemically complete treatment. Therefore, no serial biomarkers could be recorded for evaluation and prediction of cancer recurrence. In this pilot study, urinary exosomal thyroglobulin provides a non-invasive, reproducible, convenient, serial and correct follow-up for patients with thyroid cancer, because the investigators use peptide sequence to quantify the levels of thyroglobulin in urine exosome. Significant reduction in cost-spending in rhTSH consumption, and patients do not need to stop using thyroid hormone during the course of cancer follow-up. In recent years, the progress of peptides mass spectrometry provided a cost-effective, correct and new pathway for the discovery of biomarkers. Large profiling of proteomics of human urine reveled different follow-up manners. In the viewpoints of oncology, one option is to find new biomarkers for earlier diagnosis of various cancers, and the other is to make a breakthrough for follow-up residual tumor and cancer recurrence. The goal of our pilot study is trying to find the new pathway for tracking the biomarker in patients with thyroid cancer receiving ablative surgery and radioactive I-131 treatment.

ELIGIBILITY:
Inclusion Criteria:diagnosed patients with thyroid papillary, follicular and anaplastic thyroid cancer, post-operation follow up

-

Exclusion Criteria:

* Unclearly diagnosed patients with thyroid papillary, follicular and anaplastic thyroid cancer

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The investigators will enroll 150 post-operative patients with papillary, follicular or anaplastic thyroid cancer, and collect their urine samples in outpatient clinic per year. The investigators will analyze the urine exosomal proteins and probable biological markers, including thyroglobulin and galectin-3. The investigators hope to find the prognostic biological markers via this prospective study. The investigators further hope to find newly therapeutic and follow-up pathway for such patients with well-differentiated or anaplastic thyroid cancer.
Sampling Method: Probability Sample
Enrollment: 74 (Actual)
Dates: Start 2018-08-03 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2024-02-20 (Actual)

PRIMARY OUTCOMES:
Prognostic biological markers via this prospective study | 3 years
  The study was designed as prospective pattern, and the investigators enrolled thyroid cancer with follow-up, then urine exosome protein will be measured and reported. The investigators try to find the correlation of outcome ( including recurrence, lymph nodes metastasis..) together with unknown/fresh biomarkers in this study and time-dependent manner.
  Such biomarkers including thyroglobulin, galectin-3, Calprotectin A8, Calprotectin A9, TKT, Annexin II, Afamin, Keratin 8, Keratin 9, Angiopoietin-1 and TIMP will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: CHIH-YUAN WANG, Doctor, Principal Investigator — Department of Internal Medicine, National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang CY, Shih SR, Chen KY, Chung YC, Huang PJ. Long-Term Changes of Urinary Exosomal Peptide Levels After Thyroidectomy in Patients with Thyroid Cancer: A Prospective Observational Study. Int J Nanomedicine. 2024 May 23;19:4667-4677. doi: 10.2147/IJN.S458931. eCollection 2024. PMID 38803995
- [Derived] Huang TY, Wang CY, Chen KY, Huang LT. Urinary Exosomal Thyroglobulin in Thyroid Cancer Patients With Post-ablative Therapy: A New Biomarker in Thyroid Cancer. Front Endocrinol (Lausanne). 2020 Jun 16;11:382. doi: 10.3389/fendo.2020.00382. eCollection 2020. PMID 32612576